CLINICAL TRIAL: NCT02484846
Title: Impaired Vigilance, and Its Effects on Cognition and Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jamie M. Zeitzer, Ph.D., Assistant Professor, Stanford University
Organization: VA Palo Alto Health Care System (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB-20650
Record Dates: First submitted 2015-06-24; First posted 2015-06-30 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Sleep Deprivation; Feeding Behavior
MeSH Terms: conditions — Sleep Deprivation; Feeding Behavior | interventions — Time; Beds

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- 60% TIB (Experimental): Participants were to spend 60% of their normal time in bed on the night prior to the second visit.
  Interventions: Behavioral: Time in bed
- 70% TIB (Experimental): Participants were to spend 70% of their normal time in bed on the night prior to the second visit.
  Interventions: Behavioral: Time in bed
- 80% TIB (Experimental): Participants were to spend 80% of their normal time in bed on the night prior to the second visit.
  Interventions: Behavioral: Time in bed
- 90% TIB (Experimental): Participants were to spend 90% of their normal time in bed on the night prior to the second visit.
  Interventions: Behavioral: Time in bed
- 100% TIB (Active Comparator): Participants were to spend 100% of their normal time in bed (i.e., no change) on the night prior to the second visit.
  Interventions: Behavioral: Time in bed
- 115% TIB (Experimental): Participants were to spend 115% of their normal time in bed on the night prior to the second visit.
  Interventions: Behavioral: Time in bed
- 130% TIB (Experimental): Participants were to spend 130% of their normal time in bed on the night prior to the second visit.
  Interventions: Behavioral: Time in bed

INTERVENTIONS:
Behavioral: Time in bed — Habitual time spent in bed for the purpose of sleep was determined at baseline. This was used to calculated the experimental time in bed the subject was to spent on the one night prior to the second lab visit.

SUMMARY:
Fifty healthy, young participants (10 male, 40 female) completed two 3-hour study sessions that were at least five days apart. The first session was a baseline. The sleep intervention took place on the night prior to Session 2, where the amount of time in bed was manipulated to be 60-130% of the individual's habitual sleep time. Within both sessions, subjective (Stanford Sleepiness Scale, SSS) and objective (Psychomotor Vigilance Test, PVT) alertness were measured. During the middle of each session, a 40-minute ad libitum meal opportunity allowed participants to eat from eight different food items. Food healthfulness, caloric density, distribution and number of calories were measured and compared to alertness levels.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-45 years
* BMI: 20-29 kg/m²
* Eat breakfast at least 5 days per week
* Wake time occurs between 5&10AM at least 5 days per week
* Time in bed for sleep between 5&10 hours at least 5 days per week

Exclusion Criteria:

* Dietary restrictions that prohibit them from selecting one of the food choices offered in the study (e.g., gluten allergies, diabetes, vegan diet, dairy avoidance, allergies to the respective food choices available),
* are currently on a calorie-restricted diet, or
* are currently at a weight that is less than 20% of their highest weight within the last three years.
* Participation in shift work within 7 nights of the experiment
* Diagnosed as having severe sleep apnea syndrome, narcolepsy or chronic insomnia
* Diagnosed as having an eating disorder
* Active serious health condition
* Regularly taking vigilance-related medication (e.g., ADHD prescribed medication)
* Typically consume more than 600 mg of coffee or more than 10 cigarettes per day

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2011-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Total calories consumed | 45 minutes
  Total calories consumed during a 45 minute meal opportunity during the each of the two study sessions.

SECONDARY OUTCOMES:
Alertness | 15 minutes
  Objective alertness was determined during each of the two study sessions during a 15 minute test of sustained attention (Psychomotor Vigilance Task).

REFERENCES:
- [Derived] Pardi D, Buman M, Black J, Lammers GJ, Zeitzer JM. Eating Decisions Based on Alertness Levels After a Single Night of Sleep Manipulation: A Randomized Clinical Trial. Sleep. 2017 Feb 1;40(2). doi: 10.1093/sleep/zsw039. PMID 28364494